CLINICAL TRIAL: NCT02202837
Title: Defining Which Remission Criterion At Month 6 Predicts Remission At Month 12 In A Real Life Clinical Practice, In A Cohort Of Rheumatoid Arthritis Patients Treated With Etanercept (Enbrel (Registered))
Brief Title: Study With Etanercept Focusing on Remission and Predictability of Remission in Real Life Clinical Practice
Acronym: REACH RA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801378; B1801378 (Other: Alias Study Number); REACH-RA (Other: Alias Study Number)
Record Dates: First submitted 2014-07-15; First posted 2014-07-29 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Etanercept First: Adult patients with RA who receive etanercept as first biologic, according to prevailing Belgian reimbursement criteria
  Interventions: Drug: etanercept
- Etanercept second: Adult patients who receive etanercept as second biologic, according to prevailing Belgian reimbursement criteria
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — etanercept 1 x 50 mg/week or 2 x 25mg/week
  Groups: Etanercept First
Drug: etanercept — etanercept 1 x 50 mg/week or 2 x 25mg/week
  Groups: Etanercept second

SUMMARY:
Defining Which Remission Criterion at Month 6 Predicts Remission at Month 12 in a Real Life Clinical Practice, in a Cohort of Rheumatoid Arthritis Patients Treated with Etanercept

DETAILED DESCRIPTION:
The analysis of the primary endpoint will be based on a logistic regression defining the dependent variable as the remission at Month 12 and the 5 independent variables as CDAI, SDAI, DAS28, DAS28 and Ultrasound, and EULAR Boolean definition for clinical practice and clinical studies.

This analysis will be conducted in each arm of the study as well as after a pooling of both patient groups.

In this context it seems reasonable to ensure the completion of the study by a total approximate number of 100 patients (approximately 50 patients per arm). In order to ensure 50 completers in each arm, 70 patients will be recruited at baseline, taking into account a drop out rate of 30% over 1 year period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active RA who start treatment with etanercept according to the prevailing reimbursement criteria and dosing in line with the SmPC.

   1. First cohort: Etanercept is the first biological product prescribed.
   2. Second cohort: Etanercept is the second biological product prescribed.
2. Capable of understanding and willing to provide signed and dated written, voluntary informed consent before any protocol-specific procedures are performed.
3. Eighteen (18) years of age or older at time of consent.

Exclusion Criteria:

1. History of or current psychiatric illness that would interfere with the subject's ability to comply with protocol requirements or to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with moderate-to-severe RA in daily clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Belgium (35):
  - CHU Dinant Godinne, Yvoir, Namur
  - ASZ Aalst, Aalst
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - St. Lucas ZH, Assebroeck
  - St-Lucas Ziekenhuis, Assebroek
  - Centre Hospitalier Universitarie Brugmann, Brussels
  - CHIREC, Brussels
  - Private Practice, Champion
  - AZ Sint Blasius, Dendermonde
  - AZ Alma, Eeklo
  - Biomedical Research Institute/ Department of Rheumatology, Genk
  - Private Practice Rheumatology, Genk
  - ReumaClinic, Genk
  - Reumatologie Associatie, Genk
  - Private Practice, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - GHdC, Gilly
  - Private Practice, Grand-Manil
  - AZ Groeninge Campus Sint Maarten, Kortrijk
  - CHU Tivoli, La Louvière
  - Centre Hospitalier Universitaire Sart Tilman, Department of Rheumatology, Liège
  - CHU Sart Tilman/ Department of Rheumatology, Liège
  - CHU, Liège
  - Louisastraat 18, Mechelen
  - CHU Ambroise Pare, Mons
  - Hôpital Saintethérèse, Montigny Sur Sambre
  - ISPPC de Charleroi, Montigny-le-Tilleul
  - AZ Damiaan, Ostend
  - Office of Maenaut Kristien, Schoten
  - Sint-Andries Ziekenhuis, Tielt
  - CH Peltzer-Tourelle, Verviers
  - Avenue G Therasse 1, Yvoir
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801378&StudyName=Study%20with%20Etanercept%20focusing%20on%20remission%20and%20predictability%20of%20remission%20in%20real%20life%20clinical%20practice

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: First Intention: Participants with rheumatoid arthritis (RA) who received Etanercept as their first biological product, according to prevailing reimbursement criteria in Belgium were observed prospectively for 12 months. The dose and frequency of drug was decided by physician based on Summary of Product Characteristics (SmPC).
- Etanercept: Second Intention: Participants with RA who received Etanercept as second biological product (either after use of another anti-TNF or another mechanism of action), according to prevailing reimbursement criteria in Belgium were observed prospectively for 12 months. The dose and frequency of drug was decided by physician based on SmPC.
Period: Overall Study
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Started | 140 | 17
Completed | 87 | 12
Not Completed | 53 | 5
Not completed — Enbrel treatment discontinued | 36 | 4
Not completed — Other | 10 | 0
Not completed — Lost to Follow-up | 7 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis set (BAS) consisted of all participants enrolled in the study who were seen at baseline, whether from first or second cohort.
Groups:
- Etanercept: First Intention: Participants with RA who received Etanercept as their first biological product, according to prevailing reimbursement criteria in Belgium were observed prospectively for 12 months. The dose and frequency of drug was decided by physician based on SmPC.
- Total: Total of all reporting groups
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention | Total
Number analyzed (Participants) | 140 | 17 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.21 (13.55) | 56.16 (11.63) | 56.21 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 11 | 104
  Male | 47 | 6 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Activity Score Based on 28-Joints Count (DAS28) Less Than (<) 2.6 at Month 6 and Maintained Till Month 12
Description: DAS28 was a measure of disease activity in participants with rheumatoid arthritis. DAS28 was calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joints count, C-reactive protein (CRP) (milligrams per liter [mg/L]) or erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) levels and patient global assessment (PGA) of disease activity on a 0-100 mm scale (scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicated worst health condition). DAS28 score range from 0 (none) to 9.4 (extreme disease activity). DAS28 [less than or equal to] <=3.2 implied low disease activity and greater than (>) 3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28 less than (<) 2.6 implied remission.
Time Frame: Month 6 up to Month 12
Population: The completers analysis data set (CAS) consisted of all participants enrolled in study and who completed 12-month study, whether or not they missed some follow-up visits and regardless of cohort (first or second intention). Here, "N" (number of participants analyzed) signifies participants who were evaluable for this specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 76 | 10
percentage of participants | 43.4 [32.1 to 55.3] | 30.0 [6.67 to 65.3]

2. Primary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Less Than or Equal to (<=) 3.3 at Month 6 and Maintained Till Month 12
Description: The SDAI was the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, physician (evaluator) global assessment of disease (EGA) and PGA (assessed on a 0 mm [very well] to 10 mm [extremely bad] scale; higher scores indicated worst health condition) and CRP (mg/dL). SDAI total score ranged from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. SDAI >3.4 to 11 implied low disease activity, >11 to 26 implied moderate disease activity, >26 implied high disease activity and <=3.3 implied disease remission.
Time Frame: Month 6 up to Month 12
Population: The CAS consisted of all participants enrolled in the study and who completed the 12-month study, whether or not they missed some follow-up visits and regardless of the cohort (first or second intention). Here, "N" signifies those participants who were evaluable for this specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 73 | 9
percentage of participants | 13.7 [6.77 to 23.8] | 22.2 [2.81 to 60.0]

3. Primary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) <=2.8 at Month 6 and Maintained Till Month 12
Description: The CDAI was the numerical sum of four outcome parameters: TJC and SJC based on a 28-joint assessment, EGA and PGA (assessed on a 0 mm [very well] to 10 mm [extremely bad] scale; higher scores indicated worst health condition). CDAI total score ranged from 0-76 with higher scores indicating increased disease activity.
Time Frame: Month 6 up to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 78 | 11
percentage of participants | 3.85 [0.80 to 10.8] | 18.2 [2.28 to 51.8]

4. Primary Outcome: Percentage of Participants With Remission at Month 6 and Maintained Till Month 12 Based on American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) (Clinical Studies) Boolean Criterion
Description: The ACR/EULAR Boolean-based remission rate measured the severity of disease. A participant was considered as having achieved the Boolean-based ACR/EULAR remission at a visit if all of the following 4 criteria were met at that visit: TJC (in 28 joints) <=1; SJC (in 28 joints) <=1; CRP<=1 mg/dl; PGA<=1 (assessed on a 0 mm [very well] to 10 mm [extremely bad] scale; higher scores indicated worst health condition).
Time Frame: Month 6 up to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 74 | 9
percentage of participants | 2.70 [0.33 to 9.42] | 0 [0 to 33.6]

5. Primary Outcome: Percentage of Participants With Remission at Month 6 and Maintained Till Month 12 Based on American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) (Clinical Practice) Boolean Criterion
Description: The ACR/EULAR Boolean-based remission rate measured the severity of disease. A participant was considered as having achieved the Boolean-based ACR/EULAR remission at a visit if all of the following 4 criteria were met at that visit: TJC (in 28 joints) <=1; SJC (in 28 joints) <=1 and PGA<=1 (assessed on a 0 mm [very well] to 10 mm [extremely bad] scale; higher scores indicated worst health condition).
Time Frame: Month 6 up to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 79 | 11
percentage of participants | 11.4 [5.34 to 20.5] | 18.2 [2.28 to 51.8]

6. Primary Outcome: Percentage of Participants With Remission Based on Seven-Joint Ultrasound (US7) Measurements at Month 6 and Maintained Till Month 12
Description: A participant was in remission based on US7: if US7 synovitis sum score in grey-scale Ultrasonography (GSUS) =0, Power Doppler Ultrasonography (PDUS) =0 and erosion sum score in GSUS=0. US7 score is musculoskeletal ultrasonography (MKUS) composite scoring system which combined soft tissue lesions (synovitis) and destructive processes (erosions) in a single scoring system. US7 score included MKUS examination of the following joints of the more clinically affected side: wrist, metacarpophalangeal (MCP) II and III, proximal interphalangeal (PIP) II and III, metatarsophalangeal (MTP) II and V. The joints were examined by GSUS and PDUS for synovitis. Synovitis in GSUS and PDUS was analyzed on a scale of 0-3 (GSUS: 0=no synovitis, 3=severe synovitis; higher score=more synovitis); (PDUS: 0=no intraarticular color signal, 3 = >=50% of the intraarticular area filled with color signals). Erosions in GSUS and PDUS were calculated on a binary basis 0 and 1 where 0=no remission and remission=1.
Time Frame: Month 6 up to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 2
percentage of participants | 0 [0 to 70.8] | 0 [0 to 84.2]

7. Primary Outcome: Percentage of Participants With Remission Based on Disease Activity Score Based on 28-Joints Count (DAS28) in Combination With Seven-Joint Ultrasound (US7) Measurement at Month 6 and Maintained Till Month 12
Description: Remission based on DAS28 + US7: DAS28 <2.6 and US7 synovitis sum score in GSUS=0, PDUS=0 and US7 erosion sum score in GSUS=0. DAS28: SJC + TJC in 28 joints count + CRP(mg/L) or ESR(mm/hr) levels and PGA on 0-100 mm scale (0 mm [very well] to 100 mm [extremely bad], higher scores indicated worst health condition). U7 Remission: US7 synovitis sum score in GSUS=0, PDUS=0 and erosion sum score in GSUS=0. US7 score is MKUS composite scoring system which combined soft tissue lesions(synovitis) and destructive processes(erosions) in single scoring system. US7 score included MKUS examination of given joints: wrist, MCP II and III, PIP II and III, MTP II and V. Joints were examined by GSUS and PDUS for synovitis on scale of 0-3 (GSUS: 0=no synovitis, 3=severe synovitis; higher score=more synovitis); (PDUS: 0=no intraarticular color signal, 3 = >=50% of intraarticular area filled with color signals). Erosions in GSUS and PDUS were calculated on binary basis 0 (no remission) and 1 (remission).
Time Frame: Month 6 up to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 2
percentage of participants | 0 [0 to 70.8] | 0 [0 to 84.2]

8. Secondary Outcome: Percentage of Participants With Disease Activity Score Based on 28-Joints Count (DAS28) <2.6 at Month 3, 6, 9 and 12
Description: DAS28 was a measure of disease activity in participants with rheumatoid arthritis. DAS28 was calculated from SJC and TJC using 28 joints count, CRP (mg/L) or ESR) (mm/hr) levels and PGA of disease activity on a 0-100 mm scale (scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicated worst health condition). DAS28 score range from 0 (none) to 9.4 (extreme disease activity). DAS28 <=3.2 implied low disease activity and > 3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28 <2.6 implied remission.
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 86 | 12
percentage of participants
  Month 3: number analyzed (Participants) | 56 | 9
  Month 3 | 50.0 [36.3 to 63.7] | 33.3 [7.49 to 70.1]
  Month 6: number analyzed (Participants) | 76 | 10
  Month 6 | 56.6 [44.7 to 67.9] | 60.0 [26.2 to 87.8]
  Month 9: number analyzed (Participants) | 53 | 7
  Month 9 | 50.9 [36.8 to 64.9] | 28.6 [3.67 to 71.0]
  Month 12: number analyzed (Participants) | 76 | 10
  Month 12 | 51.3 [39.6 to 63.0] | 40.0 [12.2 to 73.8]

9. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) <=3.3 at Month 3, 6, 9 and 12
Description: The SDAI was the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, EGA and PGA (assessed on a 0 mm [very well] to 10 mm [extremely bad] scale; higher scores indicated worst health condition) and CRP (mg/dL). SDAI total score ranged from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. SDAI >3.4 to 11 implied low disease activity, >11 to 26 implied moderate disease activity, >26 implied high disease activity and <=3.3 implied disease remission.
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 84 | 12
percentage of participants
  Month 3: number analyzed (Participants) | 55 | 8
  Month 3 | 12.7 [5.27 to 24.5] | 12.5 [0.32 to 52.7]
  Month 6: number analyzed (Participants) | 73 | 9
  Month 6 | 19.2 [10.9 to 30.1] | 44.4 [13.7 to 78.8]
  Month 9: number analyzed (Participants) | 50 | 7
  Month 9 | 28.0 [16.2 to 42.5] | 14.3 [0.36 to 57.9]
  Month 12: number analyzed (Participants) | 69 | 9
  Month 12 | 17.4 [9.32 to 28.4] | 11.1 [0.28 to 48.3]

10. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) <=2.8 at Month 3, 6, 9 and 12
Description: as for outcome 3
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 86 | 12
percentage of participants
  Month 3: number analyzed (Participants) | 65 | 11
  Month 3 | 12.3 [5.47 to 22.8] | 18.2 [2.28 to 51.8]
  Month 6: number analyzed (Participants) | 78 | 11
  Month 6 | 7.69 [2.88 to 16.0] | 36.4 [10.9 to 69.2]
  Month 9: number analyzed (Participants) | 56 | 8
  Month 9 | 23.2 [13.0 to 36.4] | 0.00 [0.00 to 36.9]
  Month 12: number analyzed (Participants) | 75 | 10
  Month 12 | 14.7 [7.56 to 24.7] | 10.0 [0.25 to 44.5]

11. Secondary Outcome: Percentage of Participants With Remission Based on American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) (Clinical Studies) Boolean Criterion at Month 3, 6, 9 and 12
Description: as for outcome 4
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 85 | 12
percentage of participants
  Month 3: number analyzed (Participants) | 56 | 9
  Month 3 | 5.36 [1.12 to 14.9] | 11.1 [0.28 to 48.3]
  Month 6: number analyzed (Participants) | 74 | 9
  Month 6 | 6.76 [2.23 to 15.1] | 11.1 [0.28 to 48.3]
  Month 9: number analyzed (Participants) | 51 | 7
  Month 9 | 5.88 [1.23 to 16.2] | 0.00 [0.00 to 41.0]
  Month 12: number analyzed (Participants) | 73 | 10
  Month 12 | 9.59 [3.94 to 18.8] | 0.00 [0.00 to 30.9]

12. Secondary Outcome: Percentage of Participants With Remission Based on American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) (Clinical Practice) Boolean Criterion at Month 3, 6, 9 and 12
Description: as for outcome 5
Time Frame: Month 3, 6, 9 and 12
Population: The CAS consisted of all participants enrolled in the study and who completed the 12-month study, whether or not they missed some follow-up visits and regardless of the cohort (first or second intention).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 87 | 12
percentage of participants
  Month 3: number analyzed (Participants) | 66 | 12
  Month 3 | 10.6 [4.37 to 20.6] | 16.7 [2.09 to 48.4]
  Month 6: number analyzed (Participants) | 79 | 11
  Month 6 | 16.5 [9.06 to 26.5] | 45.5 [16.8 to 76.6]
  Month 9: number analyzed (Participants) | 57 | 8
  Month 9 | 26.3 [15.5 to 39.7] | 25.0 [3.19 to 65.1]
  Month 12: number analyzed (Participants) | 80 | 11
  Month 12 | 18.8 [10.9 to 29.0] | 18.2 [2.28 to 51.8]

13. Secondary Outcome: Percentage of Participants With no Signs of Ultrasound Synovitis (Ultrasound Remission) at Month 6 and 12
Description: A participant was in remission based on US7: if US7 synovitis sum score in GSUS =0, PDUS =0 and erosion sum score in GSUS=0. US7 score is MKUS composite scoring system which combined soft tissue lesions (synovitis) and destructive processes (erosions) in a single scoring system. US7 score included MKUS examination of the following joints of the more clinically affected side: wrist, MCP II and III, PIP II and III, MTP II and V. The joints were examined by GSUS and PDUS for synovitis. Synovitis in GSUS and PDUS was analyzed on a scale of 0-3 (GSUS: 0=no synovitis, 3=severe synovitis; higher score=more synovitis); (PDUS: 0=no intraarticular color signal, 3 = >=50% of the intraarticular area filled with color signals). Erosions in GSUS and PDUS were calculated on a binary basis 0 and 1 where 0=no remission and remission=1.
Time Frame: Month 6 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 2
percentage of participants
  Month 6 | 0.00 [0.00 to 70.8] | 0.00 [0.00 to 70.8]
  Month 12 | 0.00 [0.00 to 70.8] | 0.00 [0.00 to 70.8]

14. Secondary Outcome: Percentage of Participants With Remission Based on Disease Activity Score Based on 28-Joints Count (DAS28) in Combination With Seven-Joint Ultrasound (US7) Measurement at Month 6 and Month 12
Description: as for outcome 7
Time Frame: Month 6 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 2
percentage of participants
  Month 6 | 0.00 [0.00 to 70.8] | 0.00 [0.00 to 84.2]
  Month 12 | 0.00 [0.00 to 70.8] | 0.00 [0.00 to 84.2]

15. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count (DAS28) at Month 6 and 12
Description: DAS28 was a measure of disease activity in participants with rheumatoid arthritis. DAS28 was calculated from SJC and TJC using 28 joints count, CRP (mg/L) or ESR (mm/hr) levels and PGA of disease activity on a 0-100 mm scale (scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicated worst health condition). DAS28 score range from 0 (none) to 9.4 (extreme disease activity). DAS28 <=3.2 implied low disease activity and > 3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28 <2.6 implied remission.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 86 | 12
units on a scale
  Baseline | 5.06 (1.15) | 5.32 (1.44)
  Change at Month 6: number analyzed (Participants) | 76 | 10
  Change at Month 6 | 2.39 (1.21) | 1.92 (2.27)
  Change at Month 12: number analyzed (Participants) | 75 | 10
  Change at Month 12 | 2.36 (1.29) | 1.37 (1.01)

16. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Month 6 and 12
Description: as for outcome 9
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 84 | 12
units on a scale
  Baseline | 32.2 (13.67) | 35.83 (19.86)
  Change at Month 6: number analyzed (Participants) | 73 | 9
  Change at Month 6 | 21.06 (11.17) | 19.62 (18.80)
  Change at Month 12: number analyzed (Participants) | 68 | 9
  Change at Month 12 | 20.30 (12.49) | 12.10 (8.29)

17. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Month 6 and 12
Description: as for outcome 3
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 86 | 12
units on a scale
  Baseline | 31.12 (13.15) | 34.17 (18.96)
  Change at Month 6: number analyzed (Participants) | 78 | 11
  Change at Month 6 | 20.06 (10.46) | 15.64 (16.64)
  Change at Month 12: number analyzed (Participants) | 75 | 10
  Change at Month 12 | 18.85 (13.04) | 13.20 (11.71)

18. Secondary Outcome: Change From Baseline in Seven-Joint Ultrasound (US7) Synovitis Grey-Scale Ultrasonography (GSUS) Score at Month 6 and 12
Description: US7 score was MKUS composite scoring system which combined soft tissue lesions (synovitis) and destructive processes (erosions) in a single scoring system. GSUS is a scoring system use to determine synovitis. The joints were examined by GSUS for synovitis from a dorsal and palmar aspect. The US7 synovitis sum score in GSUS was the sum of the scores for 9 following parts (wrist dorsal, wrist palmar, wrist ulnar, MCP 2 palmar, MCP 3 palmar, PIP 2 palmar, PIP 3 palmar, MTP 2 dorsal, MTP 5 dorsal) on a scale ranging from 0 =no synovitis to 3=severe synovitis. Total US7 GSUS score ranged from 0 (no synovitis) to 27 (severe synovitis), higher score= more synovitis.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 4 | 2
units on a scale
  Baseline | 6.21 (2.67) | 9.50 (2.12)
  Change at Month 6: number analyzed (Participants) | 3 | 2
  Change at Month 6 | 3.24 (3.95) | 8.36 (2.32)
  Change at Month 12: number analyzed (Participants) | 3 | 2
  Change at Month 12 | 3.24 (4.20) | 3.00 (1.41)

19. Secondary Outcome: Change From Baseline in Seven-Joint Ultrasound (US7) Synovitis Power Doppler Ultrasonography (PDUS) Score at Month 6 and 12
Description: US7 score was MKUS composite scoring system which combined soft tissue lesions (synovitis) and destructive processes (erosions) in a single scoring system. PDUS assessed the degree of synovial inflammation of the joints of both hands. The joints were examined by PDUS from a dorsal and palmar aspect. The US7 synovitis sum score in PDUS was the sum of the scores of 13 following parts (wrist dorsal, wrist palmar, wrist ulnar, MCP 2 palmar, MCP 2 dorsal, MCP 3 palmar, MCP 3 dorsal, PIP 2 palmar, PIP 2 dorsal, PIP 3 palmar, PIP 3 dorsal, MTP 2 dorsal, MTP 5 dorsal) on a scale ranging from 0=no intraarticular color signal to 3 = >=50% of the intraarticular area filled with color signals. Total US7 PSUS scores ranges from 0=no intraarticular color signal to 39 = >=50% of the intraarticular area filled with color signals; higher scores= more severe disease.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 2
units on a scale
  Baseline | 7.90 (3.76) | 6.50 (7.78)
  Change at Month 6 | 6.29 (3.87) | 5.85 (8.70)
  Change at Month 12 | 6.90 (2.81) | 0.50 (3.54)

20. Secondary Outcome: Change From Baseline in Seven-Joint Ultrasound (US7) Tenosynovitis/Paratenonitis Grey-Scale Ultrasonography (GSUS) Score at Month 6 and 12
Description: US7 score was MKUS composite scoring system which combined soft tissue lesions (synovitis and tenosynovitis/paratenonitis) and destructive processes (erosions) in a single scoring system. GSUS was a scoring system used to determine the tenosynovitis/paratenonitis. The joints were examined by GSUS from a dorsal and palmar aspect. The US7 tenosynovitis/paratenonitis sum score in GSUS was the sum of the scores for 7 following parts (wrist dorsal, wrist palmar, wrist ulnar, MCP 2 dorsal, MCP I2 palmar, MCP 3 dorsal, MCP 3 palmar) on a scale ranging from 0 =no synovitis to 1=severe synovitis. Total US7 tenosynovitis/paratenonitis GSUS score ranged from 0 (no synovitis) to 7 (severe synovitis), higher score= more synovitis.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 1
units on a scale
  Baseline | 2.00 (2.65) | 0.00
  Change at Month 6: number analyzed (Participants) | 2 | 1
  Change at Month 6 | 0.50 (0.71) | 0.00
  Change at Month 12: number analyzed (Participants) | 2 | 1
  Change at Month 12 | 0.50 (0.71) | 0.00

21. Secondary Outcome: Change From Baseline in Seven-Joint Ultrasound (US7) Tenosynovitis/Paratenonitis Power Doppler Ultrasonography (PDUS) Score at Month 6 and 12
Description: US7 score was MKUS composite scoring system which combined soft tissue lesions (synovitis and tenosynovitis/paratenonitis) and destructive processes (erosions) in a single scoring system. PDUS assessed the degree of synovial inflammation of the joints of both hands. The joints were examined by PDUS from a dorsal and palmar aspect. The US7 tenosynovitis/paratenonitis sum score in PDUS was the sum of the scores for 7 following parts (wrist dorsal, wrist palmar, wrist ulnar, MCP 2 dorsal, MCP 2 palmar, MCP 3 dorsal, MCP 3 palmar) on a scale ranging from 0 =no synovitis to 1=severe synovitis. Total US7 tenosynovitis/paratenonitis PDUS score ranged from 0 (no synovitis) to 7 (severe synovitis), higher score= more synovitis.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 1
units on a scale
  Baseline | 0.67 (1.15) | 0.00
  Change at Month 6: number analyzed (Participants) | 2 | 1
  Change at Month 6 | 1.00 (1.41) | 0.00
  Change at Month 12: number analyzed (Participants) | 2 | 1
  Change at Month 12 | 1.00 (1.41) | 0.00

22. Secondary Outcome: Change From Baseline in Seven-Joint Ultrasound (US7) Erosion Grey-Scale Ultrasonography (GSUS) Score at Month 6 and 12
Description: US7 score was MKUS composite scoring system which combined soft tissue lesions (synovitis) and destructive processes (erosions) in a single scoring system. GSUS was a scoring system used to determine the erosions. The joints were examined by GSUS for erosions from a dorsal, palmar/plantar and radial/lateral (only MCP 2 and MTP 5) aspect. The US7 erosion sum score in GSUS was the sum of the 14 following scores (MCP 2 dorsal, MCP 2 palmar, MCP 2 radial, MCP 3 dorsal, MCP 3 palmar, PIP 2 dorsal, PIP 2 palmar, PIP 3 dorsal, PIP 3 palmar, MTP 2 dorsal, MTP 2 plantar, MTP 5 dorsal, MTP 5 plantar and MTP 5 lateral) ranging from 0 to 1. Total score ranged from 0 (no erosions) to 14 (severe erosions), higher score= more erosions. The score was based on measurements made at fingers and toes and were calculated for both left and right sides, the score of the clinically most affected side.
Time Frame: Month 6 and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
Number analyzed (Participants) | 3 | 2
units on a scale
  Baseline | 0.67 (0.58) | 5.00 (1.41)
  Change at Month 6 | 0.33 (0.58) | 1.50 (2.12)
  Change at Month 12 | 0.33 (0.58) | 0.50 (0.71)

ADVERSE EVENTS:
Time Frame: From Day 1 up to 28 days after end of treatment (12 months)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Etanercept: First Intention | Etanercept: Second Intention
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/17
Serious Adverse Events (participants affected / at risk) | 5/140 | 2/17
Other Adverse Events (participants affected / at risk) | 51/140 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: First Intention (N=140) | Etanercept: Second Intention (N=17)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — This event is a gender specific event.
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pain Chest (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: First Intention (N=140) | Etanercept: Second Intention (N=17)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Injection site reaction (General disorders) | 1 | 0
Injection site erythema (General disorders) | 2 | 1
Injection site pruritus (General disorders) | 0 | 1
Injection site hypersensitivity (General disorders) | 7 | 2
Injection site pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Body tinea (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Chlamydial infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 3 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 5 | 0
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Depressive mood (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT02202837/Prot_SAP_000.pdf